CLINICAL TRIAL: NCT06702761
Title: Assessing the Prevalence and Severity of Depression Among Cardiothoracic Surgery Healthcare Workers in Baghdad Using the PHQ-9: A Cross-Sectional Study
Brief Title: Prevalence and Severity of Depression Among Cardiothoracic Surgery Healthcare Workers in Baghdad: A PHQ-9 Cross-Sectional Study
Acronym: DEPRESS/PHQ-9
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241132
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Depression Disorders
Keywords: PHQ-9; HCWs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This observational study aims to estimate the prevalence and severity of depression in HCWs in cardiothoracic surgery departments in Baghdad City, Iraq, using a self-administered PHQ-9 questionnaire. The main questions it aims to answer are:

What is the prevalence of depression among cardiothoracic surgery healthcare workers? How is the severity of depression distributed within this group? Are there specific occupational or demographic factors associated with higher levels of depression?

Participants will:

Fill out the PHQ-9 in order to measure the severity of depressive symptoms at a specific moment in time.

Demographic and occupational details such as age, gender, years of experience and position held should be taken to look for possible relationship with depression.

DETAILED DESCRIPTION:
Major depressive disorder is a prevalent, severe, and recurring mental health condition.There is a significant difference in the prevalence of major depressive disorder across various socioeconomic contexts and countries. Depression is a debilitating mental illness, severely impacting psychosocial function and quality of life.

Individuals, including healthcare workers, are at risk of developing various psychological disorders, with depression being the most prevalent. In Iraq, healthcare workers are particularly vulnerable to psychological distress due to the nature of their job. They often have to deal with heavy workloads, night shifts, and shift work, which can take a toll on their mental well-being. These occupational stress factors can lead to burnout, anxiety, sleep problems, psychiatric disorders, or even depression. It has been reported that the screening for depression among healthcare workers is on the rise. Healthcare workers and individuals who work in the healthcare industry often experience symptoms of anxiety and depression at a significant rate.

There are several tools that can be used to screen for depressive disorders. One commonly used instrument in primary care is the Patient Health Questionnaire-9 (PHQ-9), which is a brief, self-administered, and easy-to-score tool that is well-validated for detecting and monitoring changes in depression severity. and detection of this condition in large epidemiological studies As this instrument is based on DSM-IV criteria, it tends to identify cases with Major Depressive Episode (MDE) when the scores are high. Additionally, it can be utilized to evaluate the intensity of depression by distinguishing between mild to severe cases. However, it is important to note that there is mounting evidence that the cut-off points used to determine the degree of severity may differ based on various contexts.

This study addresses the mental health gap among Iraqi healthcare workers, particularly in cardiothoracic surgery, within a healthcare system strained by war, resource shortages, and heavy patient loads. Despite these challenges, few studies assess depression in this group. Findings aim to inform mental health support policies for high-stress medical fields in Iraq.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals actively working in cardiothoracic surgery departments in Baghdad, including surgeons, anesthesiologists, nurses, and support staff.
* Participants who provide informed consent for participation in the study.
* Able to complete questionnaire form.

Exclusion Criteria:

* Individuals with a previously diagnosed psychiatric condition other than depression that could confound the results.
* Incomplete or missing responses on the PHQ-9 questionnaire.
* Refusal to provide informed consent.
* Participants are currently undergoing treatment for depression or other mental health conditions.
* Healthcare workers on long-term leave or who have not actively worked in the cardiothoracic surgery department for the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study targets cardiothoracic surgical departments' health care workers in Baghdad's hospitals. This encompasses cardiothoracic surgeons, anesthetists, nurses, perfusionists, and many related personnel who mostly come into direct contact with the patients. These persons work in conditions that may trigger mental health problems, such as extended working hours, intricate processes, and acute status of patients. The participants are chosen to be at least 18 years old, with different years of experience, and diagnosed to determine the rate of depression in the mentioned specific medical line.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Depression | Data collection will occur over a 3-months period, with each participant completing the assessment at a single point during this time frame.
  Proportion of cardiothoracic surgery HCWs at Al-Kadhimiya Teaching Hospital who exhibit depressive symptoms.
Severity of Depression | Data collection will occur over a 3-months period, with each participant completing the PHQ-9 assessment at a single point during this time frame.
  The severity of depression in this study will be determined based on the scores obtained from the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 categorizes depression severity as follows: Minimal depression: Scores 0-4, indicating little to no symptoms. Mild depression: Scores 5-9, suggesting occasional symptoms that may not significantly affect daily functioning. Moderate depression: Scores 10-14, indicating more frequent symptoms that can interfere with daily life. Moderately severe depression: Scores 15-19, showing pronounced symptoms that significantly impact daily activities. Severe depression: Scores 20-27, with symptoms that are debilitating.
Patient Health Questionnaire-9 (PHQ-9) | Data collection will occur over a 3-months period, with each participant completing the PHQ-9 assessment at a single point during this time frame.
  The total score can range from 0 to 27. Higher scores indicate greater severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Yaser aamer Eisa Alhaibi, Assistant professor, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kendrick T, Dowrick C, McBride A, Howe A, Clarke P, Maisey S, Moore M, Smith PW. Management of depression in UK general practice in relation to scores on depression severity questionnaires: analysis of medical record data. BMJ. 2009 Mar 19;338:b750. doi: 10.1136/bmj.b750. PMID 19299475
- [Result] Zimmerman M, Martinez JH, Friedman M, Boerescu DA, Attiullah N, Toba C. Speaking a more consistent language when discussing severe depression: a calibration study of 3 self-report measures of depressive symptoms. J Clin Psychiatry. 2014 Feb;75(2):141-6. doi: 10.4088/JCP.13m08458. PMID 24345406
- [Result] Haddad M, Walters P, Phillips R, Tsakok J, Williams P, Mann A, Tylee A. Detecting depression in patients with coronary heart disease: a diagnostic evaluation of the PHQ-9 and HADS-D in primary care, findings from the UPBEAT-UK study. PLoS One. 2013 Oct 10;8(10):e78493. doi: 10.1371/journal.pone.0078493. eCollection 2013. PMID 24130903
- [Result] Tracy M, Morgenstern H, Zivin K, Aiello AE, Galea S. Traumatic event exposure and depression severity over time: results from a prospective cohort study in an urban area. Soc Psychiatry Psychiatr Epidemiol. 2014 Nov;49(11):1769-82. doi: 10.1007/s00127-014-0884-2. Epub 2014 May 10. PMID 24816599
- [Result] van Dooren FE, Denollet J, Verhey FR, Stehouwer CD, Sep SJ, Henry RM, Kremers SP, Dagnelie PC, Schaper NC, van der Kallen CJ, Koster A, Pouwer F, Schram MT. Psychological and personality factors in type 2 diabetes mellitus, presenting the rationale and exploratory results from The Maastricht Study, a population-based cohort study. BMC Psychiatry. 2016 Jan 27;16:17. doi: 10.1186/s12888-016-0722-z. PMID 26817600
- [Result] Michal M, Wiltink J, Lackner K, Wild PS, Zwiener I, Blettner M, Munzel T, Schulz A, Kirschner Y, Beutel ME. Association of hypertension with depression in the community: results from the Gutenberg Health Study. J Hypertens. 2013 May;31(5):893-9. doi: 10.1097/HJH.0b013e32835f5768. PMID 23449018
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Kroenke K, Spitzer RL, Williams JB, Lowe B. The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):345-59. doi: 10.1016/j.genhosppsych.2010.03.006. Epub 2010 May 7. PMID 20633738
- [Result] Moitra M, Rahman M, Collins PY, Gohar F, Weaver M, Kinuthia J, Rossler W, Petersen S, Unutzer J, Saxena S, Huang KY, Lai J, Kumar M. Mental Health Consequences for Healthcare Workers During the COVID-19 Pandemic: A Scoping Review to Draw Lessons for LMICs. Front Psychiatry. 2021 Jan 27;12:602614. doi: 10.3389/fpsyt.2021.602614. eCollection 2021. PMID 33584383
- [Result] Soltani S, Tabibzadeh A, Zakeri A, Zakeri AM, Latifi T, Shabani M, Pouremamali A, Erfani Y, Pakzad I, Malekifar P, Valizadeh R, Zandi M, Pakzad R. COVID-19 associated central nervous system manifestations, mental and neurological symptoms: a systematic review and meta-analysis. Rev Neurosci. 2021 Jan 13;32(3):351-361. doi: 10.1515/revneuro-2020-0108. Print 2021 Apr 27. PMID 33618441
- [Result] Kim K, Lee S, Choi YH. Relationship between occupational stress and depressive mood among interns and residents in a tertiary hospital, Seoul, Korea. Clin Exp Emerg Med. 2015 Jun 30;2(2):117-122. doi: 10.15441/ceem.15.002. eCollection 2015 Jun. PMID 27752582
- [Result] Hegney DG, Craigie M, Hemsworth D, Osseiran-Moisson R, Aoun S, Francis K, Drury V. Compassion satisfaction, compassion fatigue, anxiety, depression and stress in registered nurses in Australia: study 1 results. J Nurs Manag. 2014 May;22(4):506-18. doi: 10.1111/jonm.12160. Epub 2013 Nov 1. PMID 24175955
- [Result] Kessler RC, Bromet EJ. The epidemiology of depression across cultures. Annu Rev Public Health. 2013;34:119-38. doi: 10.1146/annurev-publhealth-031912-114409. PMID 23514317
- [Result] Trivedi MH. Major Depressive Disorder in Primary Care: Strategies for Identification. J Clin Psychiatry. 2020 Mar 17;81(2):UT17042BR1C. doi: 10.4088/JCP.UT17042BR1C. PMID 32220155